CLINICAL TRIAL: NCT02792062
Title: A Phase 1, Randomized, Open-label, Crossover Study to Assess Food Effect on Single Oral Dose Administration of TAK-385 Final Formulation in Premenopausal Healthy Adult Women
Brief Title: A Food Effect Study of TAK-385 Final Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TAK-385-1011; JapicCTI-163273 (Registry Identifier: JapicCTI); U1111-1183-0020 (Other: UTN)
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-11

CONDITIONS: Japanese Premenopausal Healthy Adult Women
Keywords: Drug therapy
MeSH Terms: interventions — relugolix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- TAK-385 40 mg (Group A) (Experimental): A single oral dose of TAK-385 40 milligram (mg) (one tablet) in fasted condition without breakfast in Period 1, followed by a minimum 14-day washout period between study drugs, further followed by a single oral dose of TAK-385 40 mg (one tablet) before breakfast in Period 2, followed by a minimum 14-day washout period between study drugs and further followed by a single oral dose of TAK-385 40 mg (one tablet) after breakfast in Period 3.
  Interventions: Drug: TAK-385 40 mg
- TAK-385 40 mg (Group B) (Experimental): A single oral dose of TAK-385 40 mg (one tablet) before breakfast in Period 1, followed by a minimum 14-day washout period between study drugs, further followed by a single oral dose of TAK-385 40 mg (one tablet) after breakfast in Period 2, followed by a minimum 14-day washout period between study drugs and, further followed by a single oral dose of TAK-385 40 mg (one tablet) in fasted condition without breakfast in Period 3.
  Interventions: Drug: TAK-385 40 mg
- TAK-385 40 mg (Group C) (Experimental): A single oral dose of TAK-385 40 mg (one tablet) after breakfast in Period 1, followed by a minimum 14-day washout period between study drugs, further followed by a single oral dose of TAK-385 40 mg (one tablet) in fasted condition without breakfast in Period 2, followed by a minimum 14-day washout period between study drugs and, further followed by a single oral dose of TAK-385 40 mg (one tablet) before breakfast in Period 3.
  Interventions: Drug: TAK-385 40 mg
- TAK-385 40 mg (Group D) (Experimental): A single oral dose of TAK-385 40 mg (one tablet) in fasted condition without breakfast in Period 1, followed by a minimum 14-day washout period between study drugs, further followed by a single oral dose of TAK-385 40 mg (one tablet) after breakfast in Period 2, followed by a minimum 14-day washout period between study drugs and, further followed by a single oral dose of TAK-385 40 mg (one tablet) before breakfast in Period 3.
  Interventions: Drug: TAK-385 40 mg
- TAK-385 40 mg (Group E) (Experimental): A single oral dose of TAK-385 40 mg (one tablet) before breakfast in Period 1, followed by a minimum 14-day washout period between study drugs, further followed by a single oral dose of TAK-385 40 mg (one tablet) in fasted condition without breakfast in Period 2, followed by a minimum 14-day washout period between study drugs and, further followed by a single oral dose of TAK-385 40 mg (one tablet) after breakfast in Period 3.
  Interventions: Drug: TAK-385 40 mg
- TAK-385 40 mg (Group F) (Experimental): A single oral dose of TAK-385 40 mg (one tablet) after breakfast in Period 1, followed by a minimum 14-day washout period between study drugs, further followed by a single oral dose of TAK-385 40 mg (one tablet) before breakfast in Period 2, followed by a minimum 14-day washout period between study drugs and, further followed by a single oral dose of TAK-385 40 mg (one tablet) in fasted condition without breakfast in Period 3.
  Interventions: Drug: TAK-385 40 mg

INTERVENTIONS:
Drug: TAK-385 40 mg — TAK-385 40 mg tablet

SUMMARY:
The purpose of this study is to evaluate food effects on the pharmacokinetics of a single oral dose of TAK-385 in Japanese premenopausal healthy adult women.

DETAILED DESCRIPTION:
This is a phase 1 clinical pharmacological study of TAK-385 in Japanese premenopausal healthy adult women.

Using an open-label crossover design, food effects on the pharmacokinetics and safety of TAK-385 will be evaluated in participants receiving a single oral dose of TAK-385 40 mg in fasted condition without breakfast, before breakfast, or after breakfast.

Participants determined to be eligible will be randomly assigned to one of Groups A to F prior to study medication administration in Period 1; subsequently, participants will receive one TAK-385 40 mg tablet in fasted condition without breakfast (following a minimum 10-hour overnight fast), before breakfast (30 minutes before starting breakfast), or after breakfast (30 minutes after starting breakfast) in Periods 1, 2, and 3.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written, informed consent form prior to the initiation of any study procedures.
3. The participant is a Japanese premenopausal healthy adult woman.
4. The participant is aged 20 to 45 years, inclusive, at the time of informed consent.
5. The participant weighs at least 40.0 kilogram (kg) and has a body mass index (BMI) from 18.5 to 25.0 kilogram per square meter (kg/m^2), inclusive at Screening.
6. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to routinely use adequate contraception from the time of signing the informed consent form throughout the duration of the study.
7. The participant has experienced 3 or more consecutive regular menstrual cycles prior to the time of informed consent.

Exclusion Criteria:

1. The participant has received any investigational compound within 16 weeks (112 days) prior to the first dose of study drug in Period 1.
2. The participant has received TAK-385 in a previous clinical study.
3. The participant is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (example, spouse, parent, child, sibling) or may consent under duress.
4. The participant has uncontrolled, clinically significant neurological, circulatory, pulmonary, hepatic, renal, metabolic, gastrointestinal, urinary, or endocrine disease, or other abnormality, which may impact the ability of the participant to participate in the study or potentially confound the study results.
5. The participant has a diagnosis of abnormal menstruation.
6. The participant has undiagnosable abnormal genital bleeding.
7. The participant has a known hypersensitivity or allergy to drugs.
8. The participant has a positive urine drug test result for drug abuse or positive breath alcohol test result at Screening.
9. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
10. The participant has taken any excluded medication, supplements, or food products during the time periods listed in the Prohibited Medications and Dietary Products table.
11. The participant has used oral contraceptive or sex hormone preparations (norethindrone, norethisterone, medroxyprogesterone, estrogen, or other progestins) within 8 weeks (56 days) prior to hospitalization in Period 1 (Day -1), or gonadotropin-releasing hormone (GnRH) analogues, dienogest, danazol, or aromatase inhibitors within 16 weeks (112 days) prior to hospitalization in Period 1 (Day -1) [within 20 weeks (140 days) and 28 weeks (196 days) prior to hospitalization for 1- and 3-month sustained preparations, respectively].
12. The participant is pregnant or lactating or intending to become pregnant before the time of informed consent, during the study, or within 1 month after completing in this study; or intending to donate ova during such time period.
13. The participant has evidence of current cardiovascular disease, central nervous system disease, hepatic disease, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma, hypoxemia, hypertension, thromboembolism, seizures, allergic skin rash, gastrointestinal disease (pseudomembranous colitis), or mental disorder (especially depression-like symptoms) and resultant suicide attempt. The participant has a medical history, physical examination finding, or safety laboratory test finding reasonably indicative of a disease that would contraindicate GnRH analogues, or may interfere with the conduct of the study. This includes, but is not limited to, peptic ulcer disease, seizure disorders, and cardiac arrhythmias.
14. The participant has current or recent (within 6 months) gastrointestinal disease that may influence the absorption of drugs (that is, malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent heartburn, or any surgical intervention).
15. The participant has a history of cancer.
16. The participant has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antigen/antibody, or serological reactions for syphilis at Screening.
17. The participant has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to hospitalization in Period 1 (Day -1), or is unwilling to agree to stop using these products throughout the study.
18. The participant has poor peripheral venous access.
19. The participant has undergone whole blood collection of at least 200 milliliter (mL) within 4 weeks (28 days) or at least 400 mL within 16 weeks (112 days) prior to the start of study drug administration in Period 1.
20. The participant has undergone whole blood collection of at least 400 mL in total within 52 weeks (364 days) prior to the start of study drug administration in Period 1.
21. The participant has undergone blood component collection within 2 weeks (14 days) prior to the start of study drug administration in Period 1.
22. The participant has a clinically significant abnormal electrocardiogram (ECG) at Screening or prior to study drug administration in Period 1.
23. The participant has abnormal laboratory values that suggest a clinically significant underlying disease or alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) greater than (>)1.5 the upper limits of normal at Screening or prior to study drug administration in Period 1.
24. The participant who, in the opinion of the investigator, is unlikely to comply with the protocol or is unsuitable for any other reason.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07-04 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Fukuoka, Fukuoka, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 04 July 2016 to 31 August 2016.
Pre-assignment Details: Healthy premenopausal adult female participants were enrolled and randomized in this 3 period cross over study in 1 of 6 administration sequences to receive TAK-385 40 milligram (mg) under fasted conditions without breakfast, before breakfast, or after breakfast.
Groups:
- TAK-385: Fasted+ Before Breakfast + After Breakfast: TAK-385 40 mg, tablet, orally, under fasted conditions without breakfast following a minimum 10-hour (hr) overnight fast once on Day 1 of intervention period 1, followed by a minimum 14-day washout period between study drug, further followed by TAK-385 40 mg, tablet, orally, before 30 minutes of taking breakfast once on Day 1 of intervention period 2, followed by a minimum 14-day washout period between study drug, further followed by TAK-385 40 mg, tablet, orally, after 30 minutes of taking breakfast once on Day 1 of intervention period 3.
- TAK-385: Before Breakfast+ After Breakfast + Fasted: TAK-385 40 mg, tablet, orally, before 30 minutes of taking breakfast once on Day 1 of intervention period 1, followed by a minimum 14-day washout period between study drug, further followed by TAK-385 40 mg, tablet, orally, after 30 minutes of taking breakfast once on Day 1 of intervention period 2, followed by a minimum 14-day washout period between study drug, further followed by TAK-385 40 mg, tablet, orally, under fasted conditions without breakfast following a minimum 10-hr overnight fast once on Day 1 of intervention period 3.
- TAK-385: After Breakfast+ Fasted + Before Breakfast: TAK-385 40 mg, tablet, orally, after 30 minutes of taking breakfast once on Day 1 of intervention period 1, followed by a minimum 14-day washout period between study drug, further followed by TAK-385 40 mg, tablet, orally, under fasted conditions without breakfast following a minimum 10-hr overnight fast once on Day 1 of intervention period 2, followed by a minimum 14-day washout period between study drug, further followed by TAK-385 40 mg, tablet, orally, before 30 minutes of taking breakfast once on Day 1 of intervention period 3.
- TAK-385: Fasted+ After Breakfast + Before Breakfast: TAK-385 40 mg, tablet, orally, under fasted conditions without breakfast following a minimum 10-hr overnight fast once on Day 1 of intervention period 1, followed by a minimum 14-day washout period between study drug, further followed by TAK-385 40 mg, tablet, orally, after 30 minutes of taking breakfast once on Day 1 of intervention period 2, followed by a minimum 14-day washout period between study drug, further followed by TAK-385 40 mg, tablet, orally, before 30 minutes of taking breakfast once on Day 1 of intervention period 3.
- TAK-385: Before Breakfast+ Fasted + After Breakfast: TAK-385 40 mg, tablet, orally, before 30 minutes of taking breakfast once on Day 1 of intervention period 1, followed by a minimum 14-day washout period between study drug, further followed by TAK-385 40 mg, tablet, orally, under fasted conditions without breakfast following a minimum 10-hr overnight fast once on Day 1 of intervention period 2, followed by a minimum 14-day washout period between study drug, further followed by TAK-385 40 mg, tablet, orally, after 30 minutes of taking breakfast once on Day 1 of intervention period 3.
- TAK-385: After Breakfast+ Before Breakfast + Fasted: TAK-385 40 mg, tablet, orally, after 30 minutes of taking breakfast once on Day 1 of intervention period 1, followed by a minimum 14-day washout period between study drug, further followed by TAK-385 40 mg, tablet, orally, before 30 minutes of taking breakfast once on Day 1 of intervention period 2, followed by a minimum 14-day washout period between study drug, further followed by TAK-385 40 mg, tablet, orally, under fasted conditions without breakfast following a minimum 10-hr overnight fast once on Day 1 of intervention period 3.
Period: Intervention Period 1 (6 Days)
Arm/Group | TAK-385: Fasted+ Before Breakfast + After Breakfast | TAK-385: Before Breakfast+ After Breakfast + Fasted | TAK-385: After Breakfast+ Fasted + Before Breakfast | TAK-385: Fasted+ After Breakfast + Before Breakfast | TAK-385: Before Breakfast+ Fasted + After Breakfast | TAK-385: After Breakfast+ Before Breakfast + Fasted
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (at Least 14 Days)
Arm/Group | TAK-385: Fasted+ Before Breakfast + After Breakfast | TAK-385: Before Breakfast+ After Breakfast + Fasted | TAK-385: After Breakfast+ Fasted + Before Breakfast | TAK-385: Fasted+ After Breakfast + Before Breakfast | TAK-385: Before Breakfast+ Fasted + After Breakfast | TAK-385: After Breakfast+ Before Breakfast + Fasted
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention Period 2 (6 Days)
Arm/Group | TAK-385: Fasted+ Before Breakfast + After Breakfast | TAK-385: Before Breakfast+ After Breakfast + Fasted | TAK-385: After Breakfast+ Fasted + Before Breakfast | TAK-385: Fasted+ After Breakfast + Before Breakfast | TAK-385: Before Breakfast+ Fasted + After Breakfast | TAK-385: After Breakfast+ Before Breakfast + Fasted
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (at Least 14 Days)
Arm/Group | TAK-385: Fasted+ Before Breakfast + After Breakfast | TAK-385: Before Breakfast+ After Breakfast + Fasted | TAK-385: After Breakfast+ Fasted + Before Breakfast | TAK-385: Fasted+ After Breakfast + Before Breakfast | TAK-385: Before Breakfast+ Fasted + After Breakfast | TAK-385: After Breakfast+ Before Breakfast + Fasted
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 1 | 2 | 2 | 2 | 2 | 2
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Voluntary Withdrawal | 1 | 0 | 0 | 0 | 0 | 0
Period: Intervention Period 3 (6 Days)
Arm/Group | TAK-385: Fasted+ Before Breakfast + After Breakfast | TAK-385: Before Breakfast+ After Breakfast + Fasted | TAK-385: After Breakfast+ Fasted + Before Breakfast | TAK-385: Fasted+ After Breakfast + Before Breakfast | TAK-385: Before Breakfast+ Fasted + After Breakfast | TAK-385: After Breakfast+ Before Breakfast + Fasted
Started | 1 | 2 | 2 | 2 | 2 | 2
Completed | 1 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The pharmacokinetic (PK) analysis set included all participants who received the study drug, had no major protocol violation, fulfilled the minimum protocol specifications, and had data available for the PK analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-385: Fasted+ Before Breakfast + After Breakfast | TAK-385: Before Breakfast+ After Breakfast + Fasted | TAK-385: After Breakfast+ Fasted + Before Breakfast | TAK-385: Fasted+ After Breakfast + Before Breakfast | TAK-385: Before Breakfast+ Fasted + After Breakfast | TAK-385: After Breakfast+ Before Breakfast + Fasted | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (4.95) | 25.0 (7.07) | 33.0 (12.73) | 29.0 (2.83) | 31.5 (13.44) | 23.0 (4.24) | 28.0 (7.34)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 2 | 2 | 12
Region of Enrollment [Number; unit: participants]
  Japan | 2 | 2 | 2 | 2 | 2 | 2 | 12
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 153.5 (2.12) | 160.5 (3.54) | 156.0 (4.24) | 155.0 (0.00) | 156.0 (0.00) | 155.0 (7.07) | 156.0 (3.59)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 52.45 (3.041) | 53.55 (4.031) | 47.50 (4.950) | 46.45 (0.071) | 52.95 (0.071) | 50.70 (5.940) | 50.60 (3.980)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 22.20 (0.707) | 20.75 (0.636) | 19.40 (0.990) | 19.30 (0.000) | 21.70 (0.000) | 21.00 (0.566) | 20.73 (1.213)
Smoking Classification [Count of Participants; unit: Participants]
  Never smoked | 1 | 2 | 2 | 2 | 1 | 2 | 10
  Ex-smoker | 1 | 0 | 0 | 0 | 1 | 0 | 2
Alcohol Classification [Count of Participants; unit: Participants]
  Drinks a few days per week | 2 | 0 | 0 | 0 | 1 | 1 | 4
  Drinks a few days per month | 0 | 2 | 2 | 2 | 1 | 0 | 7
  Never drinks | 0 | 0 | 0 | 0 | 0 | 1 | 1
Caffeine Consumption [Count of Participants; unit: Participants]
  Caffeine consumption | 1 | 0 | 1 | 1 | 1 | 1 | 5
  No caffeine consumption | 1 | 2 | 1 | 1 | 1 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-385
Time Frame: Day 1: Pre-dose and at multiple time points (up to 120 hrs) post-dose
Population: The PK analysis set included all participants who received the study drug, had no major protocol violation, fulfilled the minimum protocol specifications, and had data available for the PK analysis. One participant discontinued study without receiving TAK-385 after breakfast in intervention period 3.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- TAK-385 40 mg Fasted: TAK-385 40 mg, tablets, orally, under fasted conditions without breakfast following a minimum 10-hr overnight fast, once on Day 1 of either intervention period 1, 2, or 3.
- TAK-385 40 mg Before Breakfast: TAK-385 40 mg, tablets, orally, before 30 minutes of taking breakfast, once on Day 1 of either intervention period 1, 2, or 3.
- TAK-385 40 mg After Breakfast: TAK-385 40 mg, tablets, orally, after 30 minutes of taking breakfast, once on Day 1 of either intervention period 1, 2, or 3.
Arm/Group | TAK-385 40 mg Fasted | TAK-385 40 mg Before Breakfast | TAK-385 40 mg After Breakfast
Number analyzed (Participants) | 12 | 12 | 11
nanogram per milliliter (ng/mL) | 23.44 (17.822) | 29.05 (22.868) | 10.94 (9.3726)
Statistical Analysis 1: Comparison: TAK-385 40 mg Fasted vs TAK-385 40 mg Before Breakfast; Mixed effect model with natural log-transformed Cmax of unchanged TAK-385 as dependent variables, arm, treatment period and dosing condition as fixed effects, and participants as a random effect was used to calculate the difference between the dosing conditions (value before breakfast - value in fasted condition without breakfast); Test type: Superiority or Other; p = 0.659, Mixed Models Analysis; Least Square Mean Ratio (%) = 113.06, 90% CI 2-sided [70.37 to 181.67]
Statistical Analysis 2: Comparison: TAK-385 40 mg Fasted vs TAK-385 40 mg After Breakfast; Mixed effect model with natural log-transformed Cmax of unchanged TAK-385 as dependent variables, arm, treatment period and dosing condition as fixed effects, and participants as a random effect was used to calculate the difference between the dosing conditions (value after breakfast - value in fasted condition without breakfast); Test type: Superiority or Other; p = 0.012, Mixed Models Analysis; Least Square Mean Ratio (%) = 45.43, 90% CI 2-sided [27.86 to 74.07]

2. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-385
Time Frame: Day 1: Pre-dose and at multiple time points (0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, and 120hrs; up to 120 hrs) post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | TAK-385 40 mg Fasted | TAK-385 40 mg Before Breakfast | TAK-385 40 mg After Breakfast
Number analyzed (Participants) | 12 | 12 | 11
nanogram*hour per milliliter (ng*hr/mL) | 160.5 (75.187) | 139.1 (65.653) | 79.65 (33.426)
Statistical Analysis 1: Comparison: TAK-385 40 mg Fasted vs TAK-385 40 mg Before Breakfast; Mixed effect model with natural log-transformed AUC∞ of unchanged TAK-385 as dependent variables, arm, treatment period and dosing condition as fixed effects, and participants as a random effect was used to calculate the difference between the dosing conditions (value before breakfast - value in fasted condition without breakfast); Test type: Superiority or Other; p = 0.238, Mixed Models Analysis; Least Square Mean Ratio (%) = 84.28, 90% CI 2-sided [66.09 to 107.47]
Statistical Analysis 2: Comparison: TAK-385 40 mg Fasted vs TAK-385 40 mg After Breakfast; Mixed effect model with natural log-transformed AUC∞ of unchanged TAK-385 as dependent variables, arm, treatment period and dosing condition as fixed effects, and participants as a random effect was used to calculate the difference between the dosing conditions (value after breakfast - value in fasted condition without breakfast); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Square Mean Ratio (%) = 53.20, 90% CI 2-sided [41.39 to 68.37]

3. Primary Outcome: AUC(0-120): Area Under the Plasma Concentration-time Curve From Time 0 to 120 Hours Postdose for TAK-385
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-385 40 mg Fasted | TAK-385 40 mg Before Breakfast | TAK-385 40 mg After Breakfast
Number analyzed (Participants) | 12 | 12 | 11
ng*hr/mL | 149.3 (70.354) | 130.2 (61.549) | 73.25 (30.726)
Statistical Analysis 1: Comparison: TAK-385 40 mg Fasted vs TAK-385 40 mg Before Breakfast; Mixed effect model with natural log-transformed AUC(0-120) of unchanged TAK-385 as dependent variables, arm, treatment period and dosing condition as fixed effects, and participants as a random effect was used to calculate the difference between the dosing conditions (value before breakfast - value in fasted condition without breakfast); Test type: Superiority or Other; p = 0.256, Mixed Models Analysis; Least Square Mean Ratio (%) = 84.68, 90% CI 2-sided [66.23 to 108.27]
Statistical Analysis 2: Comparison: TAK-385 40 mg Fasted vs TAK-385 40 mg After Breakfast; Mixed effect model with natural log-transformed AUC(0-120) of unchanged TAK-385 as dependent variables, arm, treatment period and dosing condition as fixed effects, and participants as a random effect was used to calculate the difference between the dosing conditions (value after breakfast - value in fasted condition without breakfast); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Square Mean Ratio (%) = 52.56, 90% CI 2-sided [40.78 to 67.74]

4. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-385
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-385 40 mg Fasted | TAK-385 40 mg Before Breakfast | TAK-385 40 mg After Breakfast
Number analyzed (Participants) | 12 | 12 | 11
ng*hr/mL | 149.3 (70.354) | 130.2 (61.549) | 73.25 (30.726)
Statistical Analysis 1: Comparison: TAK-385 40 mg Fasted vs TAK-385 40 mg Before Breakfast; Mixed effect model with natural log-transformed AUClast of unchanged TAK-385 as dependent variables, arm, treatment period and dosing condition as fixed effects, and participants as a random effect was used to calculate the difference between the dosing conditions (value before breakfast - value in fasted condition without breakfast); Test type: Superiority or Other; p = 0.256, Mixed Models Analysis; Least Square Mean Ratio (%) = 84.68, 90% CI 2-sided [66.23 to 108.27]
Statistical Analysis 2: Comparison: TAK-385 40 mg Fasted vs TAK-385 40 mg After Breakfast; Mixed effect model with natural log-transformed AUClast of unchanged TAK-385 as dependent variables, arm, treatment period and dosing condition as fixed effects, and participants as a random effect was used to calculate the difference between the dosing conditions (value after breakfast - value in fasted condition without breakfast); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Square Mean Ratio (%) = 52.56, 90% CI 2-sided [40.78 to 67.74]

5. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) or Serious TEAEs.
Time Frame: Day 1 up to 12 days after the last dose of study drug (Day 41)
Population: The safety analysis set included all participants who received at least one dose of the study drug. One participant discontinued study without receiving TAK-385 after breakfast in intervention period 3.
Measure: Number; unit: participants
Arm/Group | TAK-385 40 mg Fasted | TAK-385 40 mg Before Breakfast | TAK-385 40 mg After Breakfast
Number analyzed (Participants) | 12 | 12 | 11
participants
  TEAEs | 5 | 5 | 3
  Serious TEAEs | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With TEAEs Related to Vital Signs (Presyncope)
Time Frame: Day 1 up to 12 days after last dose of study drug (Day 41)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | TAK-385 40 mg Fasted | TAK-385 40 mg Before Breakfast | TAK-385 40 mg After Breakfast
Number analyzed (Participants) | 12 | 12 | 11
participants | 0 | 1 | 0

7. Secondary Outcome: Number of Participants With TEAEs Related to Body Weight
Time Frame: Day 1 up to 12 days after last dose of study drug (Day 41)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | TAK-385 40 mg Fasted | TAK-385 40 mg Before Breakfast | TAK-385 40 mg After Breakfast
Number analyzed (Participants) | 12 | 12 | 11
participants | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With TEAEs Related to Electrocardiograms (ECG)
Time Frame: Day 1 up to 12 days after last dose of study drug (Day 41)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | TAK-385 40 mg Fasted | TAK-385 40 mg Before Breakfast | TAK-385 40 mg After Breakfast
Number analyzed (Participants) | 12 | 12 | 11
participants | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With TEAEs Related to Clinical Laboratory Tests
Description: Clinical laboratory tests included hematology, serum chemistry, and urinalysis.
Time Frame: Day 1 up to 12 days after last dose of study drug (Day 41)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | TAK-385 40 mg Fasted | TAK-385 40 mg Before Breakfast | TAK-385 40 mg After Breakfast
Number analyzed (Participants) | 12 | 12 | 11
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 12 days (Day 41) after the last dose of study drug
Description: At each visit, investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by participant or observed by investigator was recorded, irrespective of relation to study treatment. One participant discontinued study without receiving TAK-385 after breakfast in intervention period 3.
Arm/Group | TAK-385 40 mg Fasted | TAK-385 40 mg Before Breakfast | TAK-385 40 mg After Breakfast
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 5/12 | 5/12 | 3/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-385 40 mg Fasted (N=12) | TAK-385 40 mg Before Breakfast (N=12) | TAK-385 40 mg After Breakfast (N=11)
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 3 | 3 | 1
Menstruation irregular (Reproductive system and breast disorders) | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.